CLINICAL TRIAL: NCT04002661
Title: Hypoactive Sexual Desire Disorder in Males (10-18-40-13)
Brief Title: Hypoactive Sexual Desire Disorder in Males
Acronym: HSDD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study's inclusion and exclusion criteria are tight and could not enroll any patients
Sponsor: Mohit Khera (Other)
Collaborators: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor-Investigator, Mohit Khera, Professor of Urology, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-44634
Record Dates: First submitted 2019-04-24; First posted 2019-06-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Low Libido
Keywords: Low libido; Erectile Dysfunction; Sexual desire
MeSH Terms: conditions — Erectile Dysfunction | interventions — flibanserin

STUDY DESIGN:
Intervention Model Description: Arm 1 will receive investigational product.
  Arm 2 will receive placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study medication (flibanserin 100 mg or identically matched placebo) will be provided in a randomized fashion. Randomization will be 1:1 with a block size of 4. Each individual kit will contain three bottles of 30 tablets of study medication. Each individual bottle within the kit will be labeled sequentially, for example kit 201 will include three bottles of 30 tablets labeled 201A, 201B, 201C. Kits will be numbered consecutively in the randomized order. Once a patient is confirmed eligible to participate in the study, the site will select the lowest numbered kit that has not been assigned to a subject. Subjects will be provided with the "A" bottle at their first visit. The site will mark the subject's study number on the kit and document which subject received that kit number. As subjects return for interim visits, they will be provided the "B" and "C" bottles from their previously assigned kit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Active (Active Comparator): Participants will take flibanserin 100mg orally every night for approximately 3 months.
  Interventions: Drug: Flibanserin
- Arm 2 - Placebo (Placebo Comparator): Participants will take a placebo orally every night for approximately 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Flibanserin — Flibanserin tablet
  Other Names: Addyi
  Arms: Arm 1 - Active
Drug: Placebo — Oral Tablet
  Arms: Arm 2 - Placebo

SUMMARY:
The purpose of this study is to determine if the study drug will increase sexual desire in men with HSDD. Half of the participants will take ADDYI while the other half will receive a placebo (a look-alike pill with no medicine).

DETAILED DESCRIPTION:
This pilot randomized placebo controlled study will include 60 men (30 treatment and 30 placebo). ARM 1 will take flibanserin 100mg orally every night and ARM 2 will take a placebo orally every night.

There will be four study visits and the study duration is approximately 4 months. Participants will have physicals at each visit. Blood draws for tests will be done at 3 visits and up to 4 questionnaires will completed at each visit. Study drug will randomized.

ELIGIBILITY:
Inclusion Criteria:

* Men age 18 through 69 years old
* Men who are distressed by their low libido as defined by SDI-2, and SCI-M questionnaires. (Appendices A,C)
* Men who are not depressed as defined by PHQ-9 (Patient Health Questionnaire) score of 9 or less. (Appendix D)
* Men with good erectile function as defined by IIEF greater than 22
* Men with normal testosterone and liver function values (may be on testosterone therapy)
* Men who are satisfied in their relationship or with their partners
* Men or their female partners must be willing to use one form of contraception throughout the study and 30 days after final study visit.
* Willing to give informed consent

Exclusion Criteria:

* Hypogonadal patients (less than 350 ng/dL)
* IIEF-EF less than 22
* CYP3A4 and CYP2C19 inhibitors Use of moderate or strong CYP3A4 inhibitors is prohibited for the duration of the trial, and if such medication becomes necessary, flibanserin treatment must be suspended until 2 weeks after the last dose of the CYP3A4 inhibitor
* Hepatic impairment not greater than 1.5 upper limit of normal of AST/ALT
* Men with normal to high libido
* Depressed patients as assessed by the PHQ-9 questionnaire as defined as 10 or greater.
* Men who are stressed or fatigued as determined by the PI
* Men with partners who have low libido as determined by the PI
* Men with pre-existing conditions that might predispose to hypertension
* Men who are not willing to meet the requirements for drinking alcohol during their participation in the study
* Men who are taking digoxin

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men who have a low libido defined by the SDI-2 (Sexual Desires Index-2), and SCI-M (Sexual Conerns Inventory - Male) questionnaires.
Enrollment: 8 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-01-23 (Actual)

PRIMARY OUTCOMES:
Sexual Desires Inventory-2 (SDI-2) | 3 months
  Range 2-10: Number of Participants with a significant change of at least 2 points higher than at screening.
Patient Health Questionnaire (PHQ-9) | 3 months
  Number of Participant with a significant change of at least 2 points on the PHQ-2 questionnaire after 3 months

SECONDARY OUTCOMES:
Erectile Function Change | 3 months
  Number of Participants with a significant change in erectile function and orgasmic scores of at least 2 points on the International Index of Erectile Function (Questions 2, 11, and 12) domain is considered to be 2 points higher than at screening
Sexual Concerns Inventory - Male (SCI-M) questionnaire | 3 months
  Number of Participants with a significant change of at least 2 points higher than at screening.

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Khera, MD, MBA, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant date for all primary and secondary outcome measures will be made available.